CLINICAL TRIAL: NCT03580772
Title: Functional Comparison of Two Modern Designs of Total Knee Replacement - a Post-operative Comparator Gait Study Comparing Persona MC to Attune Total Knee Replacement
Brief Title: Persona MC vs Attune Total Knee Replacement Study
Acronym: PERTUNE
Status: Terminated | Type: Observational
Why Stopped: Due to ongoing issues with recruitment, it was decided it was best to terminate the study and focus resources on other priorities.
Sponsor: University of Leeds (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Hemant Pandit, Professor of Orthopaedic Surgery, University of Leeds
Other Study IDs: IRAS241978
Record Dates: First submitted 2018-06-05; First posted 2018-07-09 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee replacement; Total knee arthroplasty; Gait analysis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Persona TKR: Patients will have undergone a medial congruent Persona total knee replacement
  Interventions: Device: Persona TKR
- Attune TKR: Patients will have undergone a Attune total knee replacement
  Interventions: Device: Attune TKR
- Control participants: Patients will not have recieved a primary TKR

INTERVENTIONS:
Device: Persona TKR — Persona® TKR (Zimmer Biomet)
  Groups: Persona TKR
Device: Attune TKR — Attune® TKR (Depuy synthes)
  Groups: Attune TKR

SUMMARY:
This study aims to compare clinical and functional outcomes of a cohort of patients that have undergone a medial congruent TKR to a similar cohort of patients that have undergone a conventional TKR and a cohort of control participants. Our null hypothesis is that there will be no difference in the functional outcome (as assessed by gait analysis) between Attune and Persona MC TKR.

DETAILED DESCRIPTION:
This cross sectional, post-operative comparator gait study aims to compare the functional and patient reported outcomes of patients that have undergone a MC TKR to an age, gender, BMI, pre-operative diagnosis with satisfactory clinical outcome at one year (OKS > 34) matched cohort of patients undergone a modern generation TKR which utilises a gradually reducing radius of curvature on the femoral component with conventional polyethylene (Attune) to a TKR with gradually reducing radius of curvature on the femoral component but a medial congruent (MC) TKR design (Persona).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and above*
2. Have undergone primary total knee replacement for either:

   1. Osteoarthritis
   2. avascular necrosis of the femur or tibia
3. Report an Oxford Knee Score greater than 34, obtained from usual clinical practice. OKS above 34 represents (range 0-48, high representing good outcome) a good outcome post-surgery.
4. Independent of study participation, patients received either commercially available Zimmer Biomet Persona MC bearing or DePuy Synthes Attune knee implants implanted in accordance with product labelling
5. 1-5 years post TKR surgery
6. An adequate understanding of written and verbal information in English in order to provide informed consent and answer the study questionnaires* * Control participants will meet same inclusion criteria except no primary TKR and OKS will not be required

Exclusion Criteria:

1. History of infection in the replaced joint and/or other local/systemic infection that may affect the prosthetic joint
2. Skeletal immaturity
3. Neuropathic arthropathy
4. Osteoporosis/any loss of musculature or neuromuscular disease that compromises the affected limb
5. Severe instability secondary to the absence of collateral ligament integrity
6. Pregnancy - routine clinical practice ensures that all female patients are asked whether they are pregnant and can safely receive x-rays or surgery as per standard consent forms
7. Patient is a member of a protected population (e.g., prisoner, mentally incompetent, etc.)
8. Patient has previously received partial or total knee arthroplasty for the ipsilateral knee
9. Patients who are unable to give voluntary informed consent.
10. Patients who are unable to walk unaided (post-surgery).
11. BMI > 40

    ** Control participants will meet the same exclusion criteria as TKR patients
12. Patients who suffer with cognitive impairment such as Parkinson's or Alzheimer's disease resulting in impaired mental capacity.
13. Patients who are unable to walk unaided.
14. Patients who suffer from dizzy spells or fainting episodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential patients that have undergone either a medial congruent Persona TKR or Attune TKR will be identified by the relevant orthopaedic surgeon. Control participants will be identified from an established database.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Knee extensor moment | Average 3 years ± 2 years post-surgery
  Maximum knee extensor moment during stair descent of the operated limb

SECONDARY OUTCOMES:
Proportion of patients able to complete each gait assessment | Average 3 years ± 2 years post-surgery
  During level walking and stair ascent/descent
Gait velocity | Average 3 years ± 2 years post-surgery
  During level walking and stair ascent/descent
Stance time | Average 3 years ± 2 years post-surgery
  During level walking and stair ascent/descent
Knee flexion-extension range of motion | Average 3 years ± 2 years post-surgery
  During level walking, stair ascent/descent and sit to stand
Knee extension moments | Average 3 years ± 2 years post-surgery
  During level walking, stair ascent and sit to stand
Knee adduction moment | Average 3 years ± 2 years post-surgery
  During level walking and stair ascent/descent
Ground reaction forces | Average 3 years ± 2 years post-surgery
  During level walking and stair ascent/descent
Sit to stand time | Average 3 years ± 2 years post-surgery
  During a sit to stand task
Knee angular velocity | Average 3 years ± 2 years post-surgery
  During a sit to stand task
Total OKS | Average 3 years ± 2 years post-surgery
  Total score, OKS function subscale and OKS pain subscale
2011 Knee Society Objective Knee Score | Average 3 years ± 2 years post-surgery
  Post-operative knee function and overall health assessment
Euro-QoL 5D (EQ-5D) index | Average 3 years ± 2 years post-surgery
  Quality of life
Forgotten Joint Score | Average 3 years ± 2 years post-surgery
  The Forgotten Joint Score is a 12-item questionnaire completed by the patient to determine how aware they are of their joint in their everyday life.

OTHER OUTCOMES:
Patient demographics | Average 3 years ± 2 years post-surgery
  age at surgery (yrs), gender (male/female), BMI
Pre-operative diagnosis | Average 3 years ± 2 years post-surgery
  osteoarthritis /avascular necrosis
ASA grade | Average 3 years ± 2 years post-surgery
  1/2/3

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Pandit, MBBS, MS, Principal Investigator — University of Leeds
Locations (1):
- Chapel Allerton Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable data from those patients that have undergone the MC TKR surgery will be transferred to the research funder, who will combine this with data from another trial (POLAR) for analysis.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available at the end of the study and will be available for three years
Access Criteria: Patient identifiable information will not be shared with the funder. Other relevant information will be shared after completing the study and analysing the data